CLINICAL TRIAL: NCT06854978
Title: R3THA Rehabilitation Feasibility and Usability Study
Acronym: RETHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Kiran Karunakaran, Research Scientist, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-1258-24; 2226174 (Other Grant/Funding Number: NSF)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke (Experimental): The study will enroll up to 10 participants with stroke who will be paired with trained therapists to receive R3THA telerehabilitation. The participants with stroke will participate in 7 training sessions. The training includes hand and arm exercises.
  Interventions: Other: RETHA

INTERVENTIONS:
Other: RETHA — The study will enroll up to 10 participants with stroke who will be paired with trained therapists to receive R3THA telerehabilitation. The participants with stroke will participate in 7 training sessions. The training includes hand and arm exercises.

SUMMARY:
The purpose of this study is to assess how the Rehabilitation Technologies for Hand and Arm (R3THA) device can be used for rehabilitation of people with stroke. the study will evaluate the feasibility of R3THA as outpatient telerehabilitation administered by trained clinicians to individuals with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. must be between the ages of 20 and 80
2. must have enough movement in my arms and hands to actively interact with the video games as determined by study staff
3. must have internet access at home.
4. must be comfortable performing basic functions on a computer, such as browsing the internet.
5. must be able to sit without a loss of balance while performing activities with my arms and hands as determined by study staff.

Exclusion Criteria:

Severe muscle spasms or stiffness (spasticity) in the affected upper limb that limits movement, as determined by study staff.

2) Thinking problems or have difficulty following instructions 3) Unable to interact with an entire computer screen due to spatial neglect 4) Difficulty understanding words spoken to me (Receptive aphasia) 5) Any other disabling nervous system condition (besides stroke) that has caused residual weakness, impaired range of motion, or spasticity 6) Severe arthritis that limits hand and arm movements 7) Not independent in functional activities/mobility prior to stroke

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
System Usability Survey | 5 weeks
  System Usability Scale is a well-established standardized metric used to measure usability perception of computer interfaces and products.
Exergame Questionnaire | 5 weeks
  It is a questionnaire developed to assess qualitative performance of the device
Performance Survey | 5 weeks
  It is a qualitative questionnaire with interview aimed at gauging the feasibility of integrating R3THA into the daily routines of individual with stroke/end users.
Fugl-Meyer Assessment for Upper Extremity | 5 weeks
  A standard clinical measure to assess the level of motor impairment in individuals with stroke.
Box and Blocks Test | 5 weeks
  box and blocks test is standard measure for hand dexterity and hand-eye coordination
Action Research Arm Test | 5 weeks
  The standard assessment for functional performance in individuals with stroke
Kinematic Assessment | 5 weeks
  Kinematic assesment to measure range of motion of the hand and arm

SECONDARY OUTCOMES:
Montreal Cognitive Assessment Test (MOCA) | 1 week
  30-item question to assess cognitive impairment in people with stroke. The score ranges from 0 to maximum score of 30. Score of 30 denotes high cognitive function while 0 is low cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Karunakaran, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No